CLINICAL TRIAL: NCT03355521
Title: Effects of Nordic Walking Training on Functional, Clinical and Biomechanics Parameters in Parkinson's Disease: a Randomized Controlled Clinical Trial
Brief Title: Effects of Nordic Walking in Parkinson Disease Patients
Acronym: Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Leonardo A. Peyré-Tartaruga, Adjunct Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: emonteiro
Record Dates: First submitted 2017-11-10; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Parkinson Disease 10
Keywords: functionality; gait; kinematics; electromyographic activity; depressive symptoms; quality of life
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 10; Depression | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: Experimental: Nordic walking Experimental: Nordic walking Training The total period of training was composed by 9-week of walking with poles, two sessions per week. The cycles were divided into four microcycles composed of three training sessions. Each training session took 60 min. Nordic walking aerobics training was used during the training period. These exercises were performed alternating volume and intensity. The training session was divided into three stages: (a) stretching, joint mobility, and heating; (b) main part (FW or NW); (c) return to the calm and ultimate stretching. The participants were trained with individualized prescription according to their maximum distance. A heart rate monitor, Model FT4 attached to the chest of the xiphoid process, was used to control the progression of intensity for the training cycles ranging from 60% to 80% of heart rate reserve. Additionally, we used the Borg RPE for training intensity control, which ranged between 13 and 17 of that scale.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic walking Experimental (Experimental): Experimental: Nordic walking Training The total period of training was composed by 9-week of walking with poles, two sessions per week. The cycles were divided into four microcycles composed of three training sessions. Each training session took 60 min. Nordic walking aerobics training was used during the training period. These exercises were performed alternating volume and intensity. The training session was divided into three stages: (a) stretching, joint mobility, and heating; (b) main part (NW); (c) return to the calm and ultimate stretching.
  Interventions: Other: Nordic Walking; Other: Free Walking
- Free walking (Active Comparator): Free walking Training The total period of training was composed by 9-week of walking without poles, two sessions per week. The cycles were divided into four microcycles composed of three training sessions. Each training session took 60 min. Free walking aerobics training was used during the training period. These exercises were performed alternating volume and intensity. The training session was divided into three stages: (a) stretching, joint mobility, and heating; (b) main part (FW); (c) return to the calm and ultimate stretching.
  Interventions: Other: Nordic Walking; Other: Free Walking

INTERVENTIONS:
Other: Nordic Walking — Nordic walking Training the total period of training was composed by 9-week of walking with poles, two sessions per week. The cycles were divided into four microcycles composed of three training sessions. Each training session took 60 min. Free walking aerobics training was used during the training period. These exercises were performed alternating volume and intensity. The training session was divided into three stages: (a) stretching, joint mobility, and heating; (b) main part (FW); (c) return to the calm and ultimate stretching.
Other: Free Walking — Free walking Training The total period of training was composed by 9-week of walking without poles, two sessions per week. The cycles were divided into four microcycles composed of three training sessions. Each training session took 60 min. Free walking aerobics training was used during the training period. These exercises were performed alternating volume and intensity. The training session was divided into three stages: (a) stretching, joint mobility, and heating; (b) main part (FW); (c) return to the calm and ultimate stretching.

SUMMARY:
The aim of this study was to evaluate and compare the effects of a Nordic and free walking training program on clinical, functional and biomechanical parameters of gait, in people with PD.

Outcomes: Motor symptoms: Staging and severity of PD, balance, walking functional mobility, self-selected walking velocity, and rehabilitation index. Non-Motor symptoms: Cognitive function, depressive symptoms, and quality of life (QL). Outcomes Biomechanics: Kinematic parameters (spatiotemporal and dynamic stability of walking) and neuromuscular parameters (amplitude of the electromyography signal, initial and final activation threshold, activation time and co-contraction index, of the following muscles: Vastus Lateralis (VL), Biceps Femoris (BF), Tibialis Anterior (TA), Gastrocnemius Medialis (GM).

DETAILED DESCRIPTION:
Introduction: Changes in clinical, functional and biomechanical parameters of gait are remarkable features in Parkinson's disease (PD). Such changes are disabling for the performance of daily living activities (DLAs) as they represent a high risk of falls and impair quality of life (QL) in this population. Although exercise is recommended as an effective model of therapeutic intervention, to minimize the symptoms of this disease, little is known about the effects of Nordic walking on motor and non-motor symptoms in patients with PD. Purpose: The aim of this study was to evaluate and compare the effects of a Nordic and free walking training program on clinical, functional and biomechanical parameters of gait, in people with PD. Experimental Design: Randomized controlled clinical trial (RCT). Study Site: Physical Education School of the Federal University of Rio Grande do Sul and the Clinical Hospital of Porto Alegre, in Porto Alegre, Rio Grande do Sul, Brazil. Methods: The sample comprised 33 participants, aged above 50 years, of both sexes, with a clinical diagnosis of idiopathic PD, with the staging of 1-4 in the Hoehn and Yahr scale (H&Y). The participants received two types of intervention: Nordic walking training program (NW, n = 16) and free walking training program (FW, n = 17), during six weeks. Aiming to evaluate the effects of the training program, the participants underwent the tests in the following period: pre-training + pre-familiarization (T1); post-familiarization + pre-training (T2); post-training (T3).

ELIGIBILITY:
Inclusion Criteria: volunteers aged over 50 years, of both sexes, with a clinical diagnosis of idiopathic PD and staging between 1 and 4 in Hoehn and Yahr Scale (H&Y).

-

Exclusion Criteria:

* Show chronic pain or presence of a migraine or nausea in daily life;
* History of labyrinthitis;
* Deep Brain Stimulation (DBS);
* The frequency of training below of 75%.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Test Timed Up and Go | Change from baseline at 9 weeks
  This teste evaluate the mobility functional in three meters of self-selected speed (TUGSS) or at forced speed (TUGFS)

SECONDARY OUTCOMES:
Locomotor Rehabilitation Index | Change from baseline at 9 weeks
  The Locomotor Rehabilitation Index is a method of determining how close is the SSW compared to the Optimum Speed (Vopt).
Self-selected walking speed - SSWS | Change from baseline at 9 weeks
  This outcome will be measure in test of walking treadmill
Optimal Walking Speed (OPT) | Change from baseline at 9 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill.
Quality of life (QoL) | Change from baseline at 9 weeks
  The quality of life will be estimated using the World Health Organization Quality of Life. (WHOQOL-short domains: physical, psychological, social relationships, environment, and general quality of life) and (WHOQOL-Long domains: sensory abilities, autonomy, Past. Present and Future Activities, social participation, death and dying, intimacy, and general quality of life).
Cognitive function | Change from baseline at 9 weeks
  This outcome will be measure for Montreal Cognitive Assessment (MoCA).
Depressive symptoms | Change from baseline at 9 weeks
  This outcome will be measure for the Geriatric Depression Scale - 15 item. The scale consists of 15 dichotomous questions in which participants are asked to answer yes or no in reference to how they felt over the past week (for instance, "Do you feel that your life is empty?," Do you feel that your situation is hopeless?). Scores range from 0 to 15 with higher scores indicating more depressive symptoms.

OTHER OUTCOMES:
Motor symptoms | Change from baseline at 9 weeks
  This outcome will be evaluated using Unified Parkinson's Disease Rating Scale. This Scale the clinician-scored monitored motor evaluation. Will be to considered 30% improvement in the Part III score hasbeen applied to deﬁne "responders. The score in each item ranges from 0 to 4, and the indicates greater impairment by the disease and the minimum, normality.
  The 14 items in the motor vehicle (the numbering of which goes from 18 to 31).
Balance Dynamics | Change from baseline at 9 weeks
  This outcome will be evaluated using Berg Balance Scale (BBS). This scale assessment of the individual's balance in 14 situations, representative of activities of the day to day, such as: stand up, get up, walk, to lean forward, to move, to turn, among others. The maximum score of a being reached of 56 points and each item has an ordinal scale of five alternatives ranging from 0 to 4 points, according to the degree of difficulty.
Balance Static | Change from baseline at 9 weeks
  This outcome will be evaluated using area of center of pressure (cm), with average velocity (IN cm/s) and root mean square (RMS). Assessments using unique measurements with force plat.
Spatial Temporal Parameters | Change from baseline at 9 weeks
  This outcome is measure a composite for: stride frequency (in Hetz), stride length (in meters), swing time (in second) and contact time (in second). This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed (in kilometros/hours).
Dynamics Stability | Change from baseline at 9 weeks
  This outcome will be evaluated using the coefficient of variation (CoV) of the Spatial Temporal Parameters: stride frequency (In Hertz), stride length (in meters), swing time (in seconds) and contact time(in seconds) in of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed.
Anthropometric data | Change from baseline at 9 weeks
  This outcome is a composite for: circumferences (in cm), height (in meters), body massa (in kilograms) and body mass index - BMI (weight and height will be combined to report BMI in kg/m^2. This outcome will be measure with balance, stadiometer and anthropometric tape.
Electromyographic Parameters | Change from baseline at 9 weeks
  This outcome is measure is a composite for: mean amplitude (in milivolts), onset (in seconds), offset (in seconds) and time of the signal and co-contraction (in seconds) of the muscles: vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) This outcome will be measured through Measuring the electromyographic activation during treadmill walking tests using an electromyograph. In of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed.
Parameters of Pendular Mechanism | Change from baseline at 9 weeks
  This outcome is measure a composite for:(external, internal and total mechanical work, Wext,Wint and Wtot, respectively, Recovery. This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo A Peyré-Tartaruga, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monteiro EP, Franzoni LT, Cubillos DM, de Oliveira Fagundes A, Carvalho AR, Oliveira HB, Pantoja PD, Schuch FB, Rieder CR, Martinez FG, Peyre-Tartaruga LA. Effects of Nordic walking training on functional parameters in Parkinson's disease: a randomized controlled clinical trial. Scand J Med Sci Sports. 2017 Mar;27(3):351-358. doi: 10.1111/sms.12652. Epub 2016 Feb 2. PMID 26833853
- See also: Effects of Nordic walking training on functional parameters in Parkinson's disease: a randomized controlled clinical trial — https://www.ncbi.nlm.nih.gov/pubmed/26833853